CLINICAL TRIAL: NCT07020468
Title: A Clinical Study on the Efficacy and Safety of Oxaliplatin + Irinotecan Liposome + 5-FU/LV as Neoadjuvant Therapy for Locally Advanced Colon and Upper Rectal Cancer
Brief Title: Neoadjuvant Therapy （NALIRIFOX） for Locally Advanced Colon and Upper Rectal Cancer
Acronym: HOPE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Hao-Kai Hu, doctor, Affiliated Cancer Hospital of Shantou University Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CancerShantouUMC
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Irinotecan Liposome; Locally Advanced Colorectal Cancer and Upper Rectal Cancer.; Neoadjuvant chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxaliplatin + Irinotecan Liposome + 5-FU/LV (Experimental)
  Interventions: Drug: NALIRIFOX

INTERVENTIONS:
Drug: NALIRIFOX — The patients with Locally Advanced Colorectal Cancer and Upper Rectal Cancer will undergo neoadjuvant treatment with irinotecan liposome combined with oxaliplatin + 5-FU/LV (NALIRIFOX), with each treatment cycle lasting 2 weeks, for a total of 3-6 cycles.

SUMMARY:
The goal of this clinical trial is to evaluating the efficacy and safety of Oxaliplatin + Irinotecan Liposome + 5-FU/LV in patients with Locally Advanced Colorectal Cancer and Upper Rectal Cancer. Patients would be included as:1. Aged between 18-75 years, with no gender restrictions; 2. Biopsy pathology confirmed as advanced colon cancer and upper rectal cancer; 3. Clinical staging of T3N+ or T4Nany with initially resectable tumors; 4. No distant metastasis observed in routine chest and abdominal CT scans.

The main question it aims to answer is Major Pathological Response Rate, referring to the proportion of patients who experience a significant reduction in the size of their tumor or near-complete pathological regression after treatment, typically assessed through a biopsy or surgical resection.

Participants will be Chemotherapy administered before surgery, with 3-6 cycles of treatment, using the chemotherapy regimen of Oxaliplatin + Irinotecan Liposome + 5-FU/LV.

DETAILED DESCRIPTION:
This study is a single-center, single-arm, prospective clinical trial. A total of 57 patients are expected to be enrolled over 24 months, with a 1-year follow-up observation period. Eligible participants who meet the inclusion criteria and do not meet the exclusion criteria will receive neoadjuvant treatment with irinotecan liposome combined with oxaliplatin + 5-FU/LV (NALIRIFOX). Treatment will be administered in 2-week cycles for 3-6 cycles, and surgery will be planned for those who meet surgical criteria. For those who do not meet surgical criteria, the subsequent treatment plan will be decided by the investigator. Postoperative adjuvant therapy will be determined by the investigator based on the patient's condition. The primary endpoint is the major pathological response (MPR) rate, and secondary endpoints include pathological complete response (pCR), R0 resection rate, objective response rate (ORR), disease control rate (DCR), disease-free survival (DFS), and safety.

Patients would be included as:1. Aged between 18-75 years, with no gender restrictions; 2. Biopsy pathology confirmed as advanced colon cancer and upper rectal cancer; 3. Clinical staging of T3N+ or T4Nany with initially resectable tumors; 4. No distant metastasis observed in routine chest and abdominal CT scans.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, both male and female are eligible;
2. ECOG score of 0-1;
3. Biopsy-confirmed pathological diagnosis of advanced-stage colon cancer or upper rectal cancer;
4. Clinical staging of T3N+ or T4Nany with initially resectable disease;
5. Routine chest and abdominal CT scans show no distant metastases;
6. Bone marrow function: neutrophils (ANC) ≥1.5×10^9/L, platelets (PLT) ≥100×10^9/L, hemoglobin (Hb) ≥70g/L;
7. Liver function: ALT, AST ≤2.5×ULN (upper limit of normal); total bilirubin ≤1.5×ULN; serum albumin ≥3 g/dL;
8. Kidney function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 ml/min (calculated using Cockcroft-Gault formula);
9. For female patients and those with reproductive potential, a negative pregnancy test must be conducted ≤72 hours prior to starting the study treatment, and they must agree to avoid pregnancy during the study treatment and for 6 months after the study treatment. For male patients with reproductive potential partners, they must agree to use adequate, medically approved contraception during the last study treatment and for 90 days afterward;
10. Must be willing to undergo the neoadjuvant chemotherapy regimen in this study and sign an informed consent form.

Exclusion Criteria:

1. Patients who have had other malignant tumors within the past 5 years (except for cured and non-recurring carcinoma in situ, basal cell carcinoma of the skin, etc.);
2. Patients with active, uncontrolled bacterial, viral, or fungal infections requiring systemic treatment, defined as persistent signs/symptoms related to infection that do not improve despite appropriate antibiotics, antiviral therapy, and/or other treatments;
3. Patients with uncontrolled systemic diseases, including unstable angina, myocardial infarction, congestive heart failure, severe unstable ventricular arrhythmias, history of severe pericardial disease, and other cardiovascular diseases; uncontrolled hypertension (defined as a systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg despite standardized antihypertensive treatment), or a history of hypertensive crisis or hypertensive encephalopathy; uncontrolled diabetes (fasting blood glucose ≥10 mmol/L);
4. Patients who are known to be allergic or intolerant to the investigational drug or its excipients in this study;
5. Any clinical indicators showing contraindications for chemotherapy and surgery;
6. Patients using strong inhibitors or inducers of CYP3A4, CYP2C8, and UGT1A1, etc.;
7. Pregnant or breastfeeding women, and women of childbearing potential who refuse to use appropriate contraception during the trial;
8. Patients who have participated in other clinical trials within 4 weeks prior to enrollment;
9. Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate | 24 months

SECONDARY OUTCOMES:
Pathological complete response rate | 24 months
  The Pathological Complete Response Rate (pCR) is typically expressed as a percentage (%). It refers to the proportion of patients in whom no cancer cells are detected in the tumor tissue after treatment, as assessed by pathological evaluation, indicating a complete response.

OTHER OUTCOMES:
R0 resection rate | 24months
  R0 resection rate is expressed as a percentage (%). It refers to the proportion of patients who can undergo a surgical resection (removal of a tumor or tissue) where the margins of the resected tissue are free from cancerous cells after the intervention of Oxaliplatin + Irinotecan Liposome + 5-FU/LV.
objective response rate | 24 months
  Objective response rate (ORR)is expressed as a percentage (%). It refers to the proportion of patients whose cancer shrinks or disappears after treatment, including complete Response (CR) or partial Response (PR).ORR= Number of patients with CR+ PR /Total number of patients in the study.
disease-free survival | 24 months
  Disease-Free Survival (DFS) refers to the period during which a patient shows no evidence of the disease returning or progressing after they have received treatment. The unit of Disease-Free Survival is typically time, and it is most often measured in months or years.
Adverse Event (AE) Incidence Rate | 24 months
  The Adverse Event (AE) Incidence Rate，as assessed by CTCAE v5.0，refers to the frequency or rate at which adverse events occur in a clinical trial or patient population.AE Incidence Rate= Number of patients experiencing at least one adverse event / Total number of patients in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Muming Xv, Study Director — Affiliated Cancer Hospital of Shantou University Medical College
Locations (1):
- Cancer Hospital of Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong SJ, Moughan J, Meropol NJ, Anne PR, Kachnic LA, Rashid A, Watson JC, Mitchell EP, Pollock J, Lee RJ, Haddock M, Erickson BA, Willett CG. Efficacy endpoints of radiation therapy group protocol 0247: a randomized, phase 2 study of neoadjuvant radiation therapy plus concurrent capecitabine and irinotecan or capecitabine and oxaliplatin for patients with locally advanced rectal cancer. Int J Radiat Oncol Biol Phys. 2015 Jan 1;91(1):116-23. doi: 10.1016/j.ijrobp.2014.09.031. Epub 2014 Nov 5. PMID 25446610
- [Background] Fernandez-Martos C, Brown G, Estevan R, Salud A, Montagut C, Maurel J, Safont MJ, Aparicio J, Feliu J, Vera R, Alonso V, Gallego J, Martin M, Pera M, Sierra E, Serra J, Delgado S, Roig JV, Santos J, Pericay C. Preoperative chemotherapy in patients with intermediate-risk rectal adenocarcinoma selected by high-resolution magnetic resonance imaging: the GEMCAD 0801 Phase II Multicenter Trial. Oncologist. 2014 Oct;19(10):1042-3. doi: 10.1634/theoncologist.2014-0233. Epub 2014 Sep 10. PMID 25209376
- [Background] Conroy T, Bosset JF, Etienne PL, Rio E, Francois E, Mesgouez-Nebout N, Vendrely V, Artignan X, Bouche O, Gargot D, Boige V, Bonichon-Lamichhane N, Louvet C, Morand C, de la Fouchardiere C, Lamfichekh N, Juzyna B, Jouffroy-Zeller C, Rullier E, Marchal F, Gourgou S, Castan F, Borg C; Unicancer Gastrointestinal Group and Partenariat de Recherche en Oncologie Digestive (PRODIGE) Group. Neoadjuvant chemotherapy with FOLFIRINOX and preoperative chemoradiotherapy for patients with locally advanced rectal cancer (UNICANCER-PRODIGE 23): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2021 May;22(5):702-715. doi: 10.1016/S1470-2045(21)00079-6. Epub 2021 Apr 13. PMID 33862000
- See also: The study protocol has not been registered on other websites. The detailed protocol will be available for viewing on this website once the clinical trial registration is approved. — https://clinicaltrials.gov/